CLINICAL TRIAL: NCT00890942
Title: Efficacy of Intramuscular Naloxone 0.4mg. in Prophylaxis of Intrathecal
Brief Title: Efficacy of Intramuscular Naloxone 0.4mg. in Prophylaxis of Intrathecal Morphine Induced Pruritus After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Tachawan Jirativanont, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si146/2009
Record Dates: First submitted 2009-04-26; First posted 2009-04-30 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Morphine Adverse Reaction
Keywords: pruritus; intrathecal morphine
MeSH Terms: conditions — Pruritus | interventions — Naloxone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- naloxone (Experimental)
  Interventions: Drug: naloxone
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: naloxone — naloxone 0.4mg.(1 ml) intramuscular
  Other Names: narcan
  Arms: naloxone
Drug: normal saline — normal saline 1 ml IM
  Arms: normal saline

SUMMARY:
The purpose of this study is to determine whether intramuscular naloxone 0.4mg. is effective in prophylaxis of intrathecal morphine induced pruritus after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* patient schedule for cesarean section ASA class 1

Exclusion Criteria:

* have contraindication for spinal block
* complicated pregnancy
* have history of drug abuse during pregnancy
* obesity BMI>35kg./m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
efficacy of intrathecal naloxone 0.4mg. in prophylaxis of intrathecal morphine induced pruritus after cesarean section | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Tachawan Jirativanont, MD, Principal Investigator — Anesthesiology department ,Siriraj hopital
Locations (1):
- Anesthesiology department, Siriraj Hospital, Mahidol University, Bangkok, Thailand